CLINICAL TRIAL: NCT01161771
Title: Effects of Cataract Extraction Surgery and Limbal Relaxing Incision on Corneal Sensation and Dry Eye
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-RES-09-004
Record Dates: First submitted 2010-07-06; First posted 2010-07-14 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with cataract and corneal astigmatism: Patients with cataract(s) and corneal astigmatism who received surgical treatment (cataract extraction and limbal-relaxing incisions)
  Interventions: Procedure: Cataract Surgery and Limbal relaxing incision

INTERVENTIONS:
Procedure: Cataract Surgery and Limbal relaxing incision — Cataract extraction and limbal-relaxing incisions

SUMMARY:
This is a multicenter evaluation of the effects of the cataract extraction and limbal relaxing incisions (LRI) on corneal sensation and dry eye signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo clear corneal cataract extraction with planned limbal relaxing incision for correction of a corneal astigmatism

Exclusion Criteria:

* Uncontrolled systemic disease
* Have undergone refractive surgery or any surgery involving a limbal or corneal incision
* Use of topical cyclosporine (Restasis) within three months of baseline/randomization visit
* Temporary or permanent occlusion of the lacrimal puncta

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cataract extraction and limbal relaxing incision
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Long Island City, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Cataract and Corneal Astigmatism
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Cataract and Corneal Astigmatism
Number analyzed (Participants) | 32
Age Continuous [Median (Full Range); unit: years] | 68.29 [51.64 to 83.84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects at Month 3 With Corneal Sensitivity < 50 Millimeters (mm) at Any of the Locations Measured
Description: The percentage of subjects at month 3 with corneal sensitivity < 50 mm at any of the locations measured. Corneal sensitivity is evaluated by using a nylon filament to measure the capability of the cornea (clear front portion of the eye) to respond to touch. The longest filament length at which a minimum of the 3 out of 5 stimulus applications produce a positive response from the subject was the corneal touch threshold (sensitivity). Measurements were taken at 5 different locations in each cornea.
Time Frame: Month 3
Population: Subjects enrolled who met the inclusion criteria of having 2 limbal relaxing incisions (LRIs) during cataract extraction. Nine (9) subjects only had 1 LRI.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Patients With Cataract and Corneal Astigmatism
Number analyzed (Participants) | 23
Percentage of Subjects
  Area 1 (Center) at Month 3 | 13
  Area 2 (Center of LRI 1) at Month 3 | 13
  Area 3 (Center of LRI 2) at Month 3 | 21.7
  Area 4 (90 degrees from LRI 1) at Month 3 | 13
  Area 5 (90 degrees from LRI 2) at Month 3 | 8.7

2. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) Total Score at Month 3
Description: Change from baseline in OSDI total score at month 3. The OSDI is a 12-question survey for subjects to document their dry eye disease symptoms. The OSDI consists of a 5-point scale (0=none of the time and 4 = all of the time), with higher scores representing greater disability. The scores are totaled over the 12 questions and converted to a score of 0-100 (0=no disability and 100=complete disability). A negative number change from baseline represents an improvement.
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Patients With Cataract and Corneal Astigmatism
Number analyzed (Participants) | 23
Scores on a Scale
  Baseline | 15.739 (8.368)
  Change from Baseline at Month 3 | -9.826 (7.912)

3. Secondary Outcome: Change From Baseline in Corneal Staining at Month 3
Description: Change from baseline in corneal staining at month 3. The cornea is the transparent front part of the eye which covers the iris and pupil. Corneal staining following administration of fluorescein dye in the eye is graded using a 6-point scale (0= no staining, 5 = severe staining) over 5 areas of the clear central part of the eye for a minimum score of 0 and a maximum score of 25. The higher the grade score, the worse the dry eye condition. A positive number change from baseline represents an increase in corneal staining (worsening of dry eye).
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Patients With Cataract and Corneal Astigmatism
Number analyzed (Participants) | 23
Scores on a Scale
  Baseline | 0.652 (1.668)
  Change from Baseline at Month 3 | 0.261 (2.158)

4. Secondary Outcome: Change From Baseline in Conjunctival Staining at Month 3
Description: Change from baseline in conjunctival staining severity score at month 3. The conjunctiva is the clear membrane covering the white surface of the eye. Conjunctival staining following ocular administration of lissamine green dye was graded using a 6-point scale (0= no staining, 5= severe staining) over 6 areas of the white part of the eye for a minimum score of 0 and a maximum score of 30. The higher the score, the worse the dry eye condition. A negative number change from baseline represents a decrease in the severity of conjunctival staining (improvement)
Time Frame: Baseline, Month 3
Population: Subjects enrolled who met the inclusion criteria of having 2 limbal incisions (LRIs) during cataract extraction. Nine (9) subjects only had 1 LRI.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Patients With Cataract and Corneal Astigmatism
Number analyzed (Participants) | 23
Scores on a Scale
  Baseline | 1.087 (2.557)
  Change from Baseline at Month 3 | -0.174 (2.949)

5. Secondary Outcome: Change From Baseline in Tear Break-Up Time at Month 3
Description: Change from baseline in tear break-up time (TBUT) at month 3. TBUT is the time required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film. A short TBUT is a sign of poor tear film. A negative number change from baseline indicates a decrease in TBUT (worsening).
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Patients With Cataract and Corneal Astigmatism
Number analyzed (Participants) | 23
Seconds
  Baseline | 16.4 (12.5)
  Change from Baseline at Month 3 | -3.71 (NA) — Mean calculated without standard deviation. No other measure of dispersion was calculated.

6. Secondary Outcome: Change From Baseline in Schirmer's Test at Month 3
Description: Change from baseline in Schirmer's Test result at month 3. The Schirmer's Test measures the rate of the secretion of tears produced by the eye over 5 minutes. The results indicate the presence of dry eye (Normal = greater than or equal to 10 millimeters (mm) of tears, Dry Eye = less than 10 mm of tears). The smaller the number, the more severe the dry eye. A positive number change from baseline indicates an increase in tears (improvement).
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters of Tears
Arm/Group | Patients With Cataract and Corneal Astigmatism
Number analyzed (Participants) | 23
Millimeters of Tears
  Baseline | 11.091 (5.163)
  Change from Baseline at Month 3 | 0.909 (5.74)

ADVERSE EVENTS:
Description: Serious Adverse Events and Adverse Events were not collected.
Arm/Group | Patients With Cataract and Corneal Astigmatism
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo